CLINICAL TRIAL: NCT01111396
Title: Longitudinal Investigation of Hippocampal Function and Morphology in ALL Patients Treated With Chemotherapy: A Monocentric, Interdisciplinary Pilot Study
Brief Title: Longitudinal Investigation of Hippocampal Function and Morphology in Acute Lymphatic Leukemia (ALL) Patients Treated With Chemotherapy
Acronym: HIF-ALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Professor Alexander Storch, MD, Dresden University of Technology
Other Study IDs: EK153052009
Record Dates: First submitted 2010-03-31; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Acute Lymphatic Leukemia
Keywords: ALL; GMALL 2003; Chemotherapy; Hippocampus
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with ALL under chemotherapy: This group consists of patients with initial diagnosis of acute lymphatic leukemia (ALL), who are enrolled into the GMALL 2003 chemotherapy study. There is no change of the initial GMALL 2003 treatment protocol for the present study.

SUMMARY:
There are two regions in the adult brain that exhibit neuronal stem and progenitor cells, generating new neurons postnatally and throughout adulthood. One is the so called subventricular zone the other is the dentate gyrus of the hippocampus. Adult neurogenesis is a physiological process representing an important functional impact for certain brain areas, especially the hippocampus. The hippocampal formation plays an important role in long-term memory and spatial navigation. Inhibition of adult neurogenesis in mice by chemotherapy or radiation is followed by significant deficits in hippocampal memory functions while hippocampus-independent memory is unaffected.

Clinical trials had shown that chemotherapy and brain radiation lead to cognitive dysfunction. However, the exact mechanisms underlying this phenomenon are still unidentified.

The aim of our study is to investigate, whether the inhibition of adult neural stem cell proliferation in the hippocampus by intrathecal chemotherapy and/or cerebral radiation is responsible for treatment induced memory deficits. We will investigate patients suffering from acute lymphatic leukaemia (ALL) that receive prophylactic intrathecal chemotherapy and brain irradiation. The study represents a longitudinal investigation including a virtual "humanized" version of the morris-water-maze to test hippocampus dependent spatial memory, as well as MR-imaging for morphological (volumetry) and biochemical (spectroscopy) data.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of acute lymphatic leukaemia (ALL)
* Treatment within the German Multicenter Adult ALL (GMALL 2003) therapy study
* Age 18 to 40 years
* Eligibility for performing study procedure
* Informed consent

Exclusion Criteria:

* Neuropsychiatric disorders
* Present contraindication for MRI investigation (e.g. pacemaker)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive patients of the Department of Internal Medicine at the Dresden University of Technology hospital, who are initially diagnosed of acute lymphatic leukemia (ALL) and included into the GMALL 2003 chemotherapy study. All treatment procedures and outcome measurements of the GMALL 2003 study (most importantly also the safety outcome measures) are regularly performed in the sub population of the present sub study. Inclusion and exclusion criteria are given below.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
Hippocampal function measured with virtual water maze test | day 0
  The hippocampal function will by studies in a longitudinal manner and thus we plan to measure the water maze test performance at several time points (time frames) of the study.
Hippocampal function measured with virtual water maze test | day 9
  The hippocampal function will by studies in a longitudinal manner and thus we plan to measure the water maze test performance at several time points (time frames) of the study.
Hippocampal function measured with virtual water maze test | day 16
  The hippocampal function will by studies in a longitudinal manner and thus we plan to measure the water maze test performance at several time points (time frames) of the study.
Hippocampal function measured with virtual water maze test | day 52
  The hippocampal function will by studies in a longitudinal manner and thus we plan to measure the water maze test performance at several time points (time frames) of the study.
Hippocampal function measured with virtual water maze test | day 70
  The hippocampal function will by studies in a longitudinal manner and thus we plan to measure the water maze test performance at several time points (time frames) of the study.
Hippocampal function measured with virtual water maze test | week 36
  The hippocampal function will by studies in a longitudinal manner and thus we plan to measure the water maze test performance at several time points (time frames) of the study.

SECONDARY OUTCOMES:
Hippocampal morphology measured by MRI | day 0
Hippocampal morphology measured by MRI | day 29
Hippocampal morphology measured by MRI | day 70
Hippocampal morphology measured by MRI | week 36
Peripheral blood cell count | day 0
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | day 26
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | day 46
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | day 71
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | week 16
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | week 22
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | week 30
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood cell count | week 41
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Peripheral blood count | week 52
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Peripheral blood cell counts for estimating the chemotherapy toxicity according to WHO criteria and the minimal residual disease activity.
Bone marrow examination | day 0
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | day 26
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | day 46
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | day 71
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | week 16
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | week 22
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | week 30
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | week 41
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.
Bone marrow examination | week 52
  Since we investigate a subpopulation of the GMALL 2003 chemotherapy study, all safety measures of the GMALL 2003 study are performed in the population of the present study.
  Bone marrow examination is investigated to extimate minimal residual disease activity and chemotherapy toxicity according to WHO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Storch, MD, Principal Investigator — Technische Universität Dresden
Locations (1):
- Dresden University of Technology University Hospital, Dresden, Germany